CLINICAL TRIAL: NCT04420481
Title: Growth Hormone Treatment in Patients With Ischemic Heart Failure and Circulating Levels of NT-proBNP
Brief Title: Growth Hormone in Ischemic Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol 2003-03-26
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure, Systolic; Ischemic Heart Disease Chronic
Keywords: Heart Failure, Systolic; Ischemic Heart Disease; Growth Hormone Treatment; Insulin Growth Factor I Resistance; Hormone Disturbance
MeSH Terms: conditions — Heart Failure, Systolic; Myocardial Ischemia; Insulin-Like Growth Factor I, Resistance To; Endocrine System Diseases | interventions — Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: A 12 month study, consisting of a 9 months' double-blind, placebo-controlled randomised growth hormone treatment phase followed by a 3 months' growth hormone treatment-free period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All care providers and patients were masked with respect to the study drug during the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth hormon group (Active Comparator): A 12 month study, consisting of a 9 months growth hormone treatment phase followed by a 3 month growth hormone treatment-free period.
  Interventions: Drug: Somatropin
- Control group (Placebo Comparator): A 12 month study, consisting of a 9 month placebo treatment phase followed by a 3 month treatment-free period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Somatropin — Dose: 1,4 mg (4,2 IE) every other day Dosage: 9 month treatment period and a 3 month follow-up period Administration: One subcutaneous injection of somatropin or corresponding placebo in the thigh or abdomen given in the evening given every other day.
  Arms: Growth hormon group
Drug: Placebo — Placebo
  Arms: Control group

SUMMARY:
In a double-blind, placebo-controlled trial, we randomly assigned 37 patients (mean age 66 years; 95% male) with ischemic heart failure (HF) (ejection fraction (EF) < 40%) to a 9-month treatment with either recombinant human GH (1.4 mg every other day) or placebo, with subsequent 3-month treatment-free follow-up. The primary outcome was change in left ventricular (LV) end-systolic volume measured by cardiac magnetic resonance (CMR). Secondary outcomes comprised changes in cardiac structure and EF. Prespecified tertiary outcomes included changes in New York Heat Association (NYHA) functional class and quality of life (QoL), as well as levels of insulin-like growth factor-1 (IGF-1) and N-terminal pro-brain natriuretic peptide (NT-proBNP).

DETAILED DESCRIPTION:
TITLE: GROWTH HORMONE IN HEART FAILURE Addition of recombinant human growth hormone to standard heart failure therapy in patients with congestive heart failure due to ischaemic heart disease.

A 12 month study, consisting of a 9 month double-blind, placebo-controlled randomised growth hormone treatment phase followed by a 3 month growth hormone treatment-free period.

STUDY PHASE: III

COORDINATING CENTRE:

Endocrine Cardiac Unit (ECU) Sahlgrenska University Hospital, Sahlgrenska S-413 45 Göteborg Sweden

STUDY PRODUCT:

Somatropin, recombinant human growth hormone (rhGH), Saizen® 8 mg (24 IE).

CONTROL PRODUCT:

Placebo for Saizen®

DOSAGE OF STUDY PRODUCT:

1,4 mg (4,2 IE) every other day.

DOSAGE:

9 month treatment period and a 3 month follow-up period. ROUTE OF ADMINISTRATION One subcutaneous injection of Saizen® of study product, or corresponding placebo in the thigh or abdomen given in the evening given every other day.

STUDY DESIGN:

Double-blind (regarding treatment), parallel, placebo-controlled, randomised.

STUDY POPULATION:

Female and male patients 75 years of age or below with congestive heart failure (NYHA class II or III) due to ischemic heart disease.

NUMBER OF PATIENTs:

54 evaluable patients. MULTICENTRE: Yes. NUMBER OF CENTRES: Four

ALLOCATION OF TREATMENT:

Randomisation to treatment if all inclusion/exclusion criteria are met.

PRIMARY OBJECTIVE:

To investigate the effect of subcutaneously administered Saizen® compared with placebo on left ventricular endsystolic volume by MRI in patients with congestive heart failure due to ischaemic heart disease.

SECONDARY OBJECTIVE:

To determine the effect of Saizen® on enddiastolic volume, left ventricular mass and left ventricular ejection fraction

TERTIARY OBJECTIVES:

To determine the effect of Saizen® on change in NYHA class after 9 months of follow up.

To determine the effect of Saizen® on circulating levels of IGF-I and IGFBP-3 and to evaluate the correlation between changes in IGF-I and the respective changes in left ventricular ejection fraction, wall stress and left ventricular mass.

To evaluate the effect of Saizen® on quality of life by using two different questionnaires (Minnesota - Living with Heart Failure and Cardiac Health Profile).

To determine the effect of Saizen® on neurohormonal activation by measuring NT-proBNP

SAFETY VARIABLES:

Hospitalization, morbidity and mortality.

* Clinical events, including tendency to fluid retention, glucose intolerance, arrhythmias and worsening heart failure.
* Electrolytes, haematology, prothrombin complex, parameters for renal and hepatic function.

ADVERSE EVENTS:

Spontaneously reported from patients and asked for. To be recorded in Case Report Forms (CRFs) and on separate Adverse Event form if serious Adverse Event.

STATISTICS AND DATABASE MANAGEMENT:

Data management will be performed by Scandinavian Contract Research Institute and when clean file is declared data will be made available to the statistician for the analysis. The analysis will be performed according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Ejection fraction at rest less than 40% at the screening visit as measured by echocardiography and a left ventricular enddiastolic diameter > 32 mm/m2
* Stable, optimised therapy for heart failure for at least 4 weeks prior to randomisation including Angiotensin converting enzyme inhibitors, or if not tolerated, angiotensin II blockers and/or digitalis. If tolerated patients should receive beta-blockers for heart failure provided they have had a stable dose for at least 3 months prior to randomisation. The dose of diuretics may vary within a given dose-range considered normal for that patient as determined by the investigator.
* Written informed consent obtained

Exclusion Criteria:

* Uncontrolled hypertension, treated or not treated with a diastolic blood pressure >105 mm Hg
* Haemodynamic clinically significant primary valvular disease or significant congenital heart disease
* Hypertrophic or idiopathic dilated cardiomyopathy
* Acute pericarditis/myocarditis
* Echocardiography findings such as mobile thrombus, significant pericardial effusion and significant left ventricular aneurysm
* Symptomatic or sustained ventricular arrhythmias within the last 3 months not adequately treated with antiarrhythmic drugs or internal cardiovertor defibrillator (ICD)
* Unstable angina pectoris, or myocardial infarction within last 3 months
* percutaneous coronary intervention performed within 6 months prior to randomization
* Planned percutaneous coronary intervention, heart transplantation, other cardiac surgery or other major surgery
* Atrial fibrillation, if a frequency > 100/min or a large frequency variation, according to clinical judgment
* Diabetes mellitus, insulin treated
* Severe liver disease (alanine aminotransferase and/or alanine aminotransferase three times upper limit of normal range laboratory values)
* Severely reduced renal function (S-Creatinine above 250 micromol/l) or suspected significant renal artery stenosis
* Uncontrolled endocrine disorders
* Ongoing treatment with calcium antagonist
* Pregnancy or lactation or females of childbearing potential taking inadequate measures to prevent pregnancy
* History of or ongoing malignant disease
* Previous treatment with growth hormone
* Patients in a catabolic state
* Known drug and/or alcohol abuse
* Inability to cooperate or administer the study drug
* Patients participating in any other clinical study, within 30 days prior to screening visit and/or during this particular study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-04-28 (Actual); Primary Completion 2012-02-25 (Actual); Study Completion 2012-02-25 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular endsystolic volume | 9 months
  Measured by CMR

SECONDARY OUTCOMES:
Change in enddiastolic volume | 9 months
  Measured by CMR
Change in left ventricular mass | 9 months
  Measured by CMR
Change in left ventricular ejection fraction | 9 months
  Measured by CMR

OTHER OUTCOMES:
Change in QoL Questionnaire | 9 months
Change in NT-proBNP level | 9 months
  blood sample

IPD SHARING:
Plan to Share IPD: Yes
Data will be share upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months
Access Criteria: A researcher that can show previous scientific merits that can be validated